CLINICAL TRIAL: NCT07322406
Title: Kaempferol Absorption and Pharmacokinetics Evaluation (K.A.P.E.)
Brief Title: Kaempferol Absorption and Pharmacokinetics Evaluation
Acronym: KAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Afshin Beheshti, Professor/Director, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25100114
Record Dates: First submitted 2025-12-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: No Disease; Mitochondria Health; Longevity; Pharmacokinetics and Biological Absorption of Kaempferol in Healthy Adult; Healthy Volunteers
Keywords: Mitochondria; Kaempferol; KMP; Pharmacokinetics; Bioavailability; Absorption; Dietary supplement; Healthy volunteers; Multi-omics
MeSH Terms: interventions — kaempferol

STUDY DESIGN:
Intervention Model Description: * All enrolled participants receive the same intervention (oral Kaempferol administered as capsules over 8 days).
  * There is no placebo group, no comparator, and no randomization.
  * Outcomes (PK, safety, and multi-omics endpoints) are assessed within the same group over time using pre- and post-intervention measurements.
  * The primary goal is pharmacokinetic characterization and biological absorption, not comparative efficacy.
Masking Description: This is an open-label, single-arm pharmacokinetic and safety study in healthy volunteers. All participants and study personnel are aware of the intervention being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kaempferol Intervention Arm (Experimental): Participants in this single-arm intervention receive oral Kaempferol (KMP) administered as capsules once daily for 8 days as part of a controlled dietary regimen. All participants undergo standardized pharmacokinetic blood and urine sampling at predefined time points, along with safety monitoring and comprehensive multi-omics analyses to assess absorption, metabolism, tolerability, and biological responses to Kaempferol.
  Interventions: Dietary Supplement: Kaempferol

INTERVENTIONS:
Dietary Supplement: Kaempferol — Kaempferol (KMP) is administered orally as encapsulated doses once daily for 8 consecutive days in healthy adult participants under controlled dietary conditions. This intervention is designed specifically for intensive pharmacokinetic characterization and biological absorption assessment, incorporating high-frequency serial blood and urine sampling across multiple time points. In contrast to typical dietary supplement studies, this intervention integrates comprehensive multi-omics profiling (including transcriptomics, miRNA-seq, metabolomics, lipidomics, proteomics, and genomic analyses) to evaluate mechanistic and functional biological responses to Kaempferol exposure. Safety and tolerability are monitored throughout the intervention period.

SUMMARY:
This study is a multi-site clinical trial designed to evaluate how the body absorbs and processes Kaempferol, a naturally occurring compound found in many plant-based foods. The primary purpose of the study is to measure the pharmacokinetics and biological absorption of Kaempferol in healthy adults.

Participants will receive Kaempferol and undergo scheduled blood and urine collections over a short study period. These samples will be used to measure Kaempferol levels in the body and to assess safety and tolerability. In addition, selected biological samples will be analyzed to explore molecular changes associated with Kaempferol exposure using advanced laboratory methods.

The study will be conducted at multiple research centers in the United States using a standardized protocol to ensure consistency across sites. The information collected will help improve understanding of how Kaempferol is absorbed and metabolized in humans and will support future research and regulatory evaluation.

DETAILED DESCRIPTION:
This multi-site interventional study evaluates the pharmacokinetics and biological absorption of Kaempferol (KMP) in a U.S. population and is designed to generate human data to inform regulatory and translational planning for Kaempferol.

Kaempferol is a diet-derived flavonoid present in plant-based foods and dietary supplements. Existing evidence supporting biological activity has largely been derived from in vitro and animal studies, with limited human clinical data describing absorption, metabolism, and excretion. Preliminary nonclinical data support measurable biological activity following oral administration, including changes consistent with altered metabolic and mitochondrial function. Prior small human studies suggest tolerability but have not provided comprehensive pharmacokinetic characterization or integrated molecular profiling. The current study is intended to address these gaps using standardized procedures across multiple U.S. clinical research sites.

Participants receive oral Kaempferol administered under controlled study conditions and complete a defined schedule of clinic visits with serial biospecimen collections. Biospecimens are processed using harmonized standard operating procedures at collection sites, with centralized laboratory analyses used to reduce variability and improve data quality. Research data are maintained using coded identifiers and stored in secure systems consistent with institutional data protection requirements.

Primary endpoint: The primary endpoint is characterization of the pharmacokinetic profile of Kaempferol, including assessment of absorption, distribution, metabolism, and excretion using serial Kaempferol and metabolite measurements in blood and urine across predefined time points.

Secondary endpoints: Secondary endpoints include exploratory assessment of biological responses associated with Kaempferol exposure using multi-omics profiling (including genomics, transcriptomics, miRNA profiling, metabolomics, lipidomics, and proteomics). Secondary analyses also include integration of molecular profiling results with participant self-reported medical history using computational approaches to explore patterns associated with Kaempferol exposure and inter-individual variability in biological response. Additional secondary endpoints include evaluation of mechanistic and functional biomarker changes associated with oxidative stress, inflammation, and metabolic health in relation to Kaempferol intake.

Safety endpoints: Safety is assessed throughout the study period. Primary safety endpoints include the incidence and characterization of adverse events (AEs) and serious adverse events (SAEs), and tolerability based on participant-reported symptoms and clinical assessments. Secondary safety endpoints include clinical laboratory evaluations, including complete blood count testing, to identify potential safety signals associated with Kaempferol administration.

All study activities are conducted under institutional review board oversight. Written informed consent is obtained prior to initiation of study procedures. A limited waiver of documentation of consent may be used only for specific preparatory dietary instructions when approved by the IRB and when required by scheduling and protocol timing. Participant confidentiality is maintained through coding of data, restricted access to identifiable information, and secure storage of study records.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 70 years

* Healthy volunteers as determined by medical history and screening assessment
* Ability to understand the study procedures and provide informed consent
* Willingness and ability to comply with all study procedures, including dietary restrictions, clinic visits, blood draws, urine collection, and follow-up assessments
* Willingness to abstain from restricted foods, beverages, and supplements as specified in the study protocol during the study period

Exclusion Criteria:

* Known allergy or hypersensitivity to Kaempferol or related flavonoids
* Pregnancy or breastfeeding
* Presence of significant acute or chronic medical conditions that could increase risk or interfere with study outcomes, including but not limited to:
* Active or chronic infections
* Cancer
* Cardiovascular disease
* Neurological or neurodegenerative disorders
* Metabolic or systemic inflammatory conditions
* Use of prescription medications or supplements known to interfere with Kaempferol metabolism or pharmacokinetic assessment
* Blood donation within 8 weeks prior to study enrollment
* Participation in another interventional clinical study within a timeframe that could interfere with study results or participant safety
* Any condition or circumstance that, in the judgment of the study investigator, would make participation unsafe or compromise data integrity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Kaempferol | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The maximum observed plasma concentration of Kaempferol following oral administration, calculated from serial plasma samples collected at predefined time points.
Time to maximum plasma concentration (Tmax) of Kaempferol | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The time elapsed from oral administration of Kaempferol to the occurrence of the maximum observed plasma concentration (Cmax), determined from serial plasma sampling.
Area under the plasma concentration-time curve (AUC) of Kaempferol | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The area under the plasma concentration-time curve of Kaempferol, calculated using noncompartmental methods to quantify overall systemic exposure following oral administration.
Plasma elimination half-life (t½) of Kaempferol | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The terminal elimination half-life of Kaempferol in plasma, estimated from the terminal phase of the concentration-time curve following oral administration.
Apparent clearance of Kaempferol | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The apparent systemic clearance of Kaempferol following oral administration, calculated using standard pharmacokinetic methods based on plasma concentration data.
Urinary excretion of Kaempferol and metabolites | From dosing on Day 1 through 24 hours after the final dose (Day 8)
  The cumulative amount of Kaempferol and its metabolites excreted in urine, determined from timed urine collections following oral administration.

SECONDARY OUTCOMES:
Differential gene expression associated with Kaempferol exposure | Baseline (Day 0 or pre-dose), Day 1 (pre-dose, 3 hours post-dose, 24 hours post-dose), Day 7 (pre-dose, 3 hours post-dose, 24 hours post-dose)
  Changes in gene expression will be quantified using RNA sequencing of peripheral blood samples. Differential expression will be reported as log2 fold change with associated statistical significance (e.g., adjusted p-values or false discovery rate) comparing post-dose time points to baseline.
Changes in circulating microRNA (miRNA) expression following Kaempferol administration | Baseline (Day 0 or pre-dose), Day 1 (pre-dose, 3 hours post-dose, 24 hours post-dose), Day 7 (pre-dose, 3 hours post-dose, 24 hours post-dose)
  Circulating miRNA expression levels will be quantified using miRNA sequencing. Outcomes will be reported as normalized expression values and log2 fold changes relative to baseline, with statistical significance assessed across post-dose time points.
Changes in plasma metabolite profiles associated with Kaempferol exposure | Baseline (Day 0 or pre-dose), Day 1 (pre-dose, 3 hours post-dose, 24 hours post-dose), Day 7 (pre-dose, 3 hours post-dose, 24 hours post-dose)
  Plasma metabolite concentrations will be measured using mass spectrometry-based metabolomics. Outcomes will be reported as relative or absolute metabolite abundances, pathway-level enrichment scores, and fold changes comparing post-dose samples to baseline.
Changes in lipidomic profiles following Kaempferol administration | Baseline (Day 0 or pre-dose), Day 1 (pre-dose, 3 hours post-dose, 24 hours post-dose), Day 7 (pre-dose, 3 hours post-dose, 24 hours post-dose)
  Lipid species concentrations will be quantified using lipidomics platforms. Results will be reported as normalized lipid abundances, fold changes from baseline, and pathway-level alterations associated with lipid metabolism.
Proteomic changes associated with Kaempferol exposure | Baseline (Day 0 or pre-dose), Day 1 (pre-dose, 3 hours post-dose, 24 hours post-dose), Day 7 (pre-dose, 3 hours post-dose, 24 hours post-dose)
  Protein abundance will be quantified using mass spectrometry-based proteomics. Outcomes will be reported as normalized protein expression levels, fold changes relative to baseline, and enrichment of biological pathways associated with Kaempferol exposure.
Integrated multi-omics pathway perturbation associated with Kaempferol exposure | Baseline (Day 0 or pre-dose) through Day 8 (24 hours after final dose)
  Integrated multi-omics analyses will be used to identify biological pathways altered following Kaempferol administration. Outcomes will be reported as pathway enrichment scores and network-level changes derived from combined transcriptomic, miRNA, metabolomic, lipidomic, and proteomic data.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Beheshti, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study includes intensive pharmacokinetic and high-dimensional multi-omics data that could increase the risk of participant re-identification, even after de-identification. In addition, data sharing is subject to institutional policies, IRB restrictions, and data governance agreements that limit external distribution of individual-level data. Aggregate results and analyses will be disseminated through peer-reviewed publications and scientific presentations.